CLINICAL TRIAL: NCT02950883
Title: Saline Hypertonic in Preschoolers With Cystic Fibrosis and Lung Structure as Measured by Computed Tomography (CT)
Brief Title: Saline Hypertonic in Preschoolers + CT
Acronym: SHIP-CT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington, the Collaborative Health Studies Coordinating Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHIP002
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Hypertonic Saline; Inhaled Saline; Digestive System Diseases; Genetic Diseases, Inborn; Lung Diseases; Pancreatic Diseases; Pathologic Processes; Respiratory Tract Diseases; Computed Tomography (CT)
MeSH Terms: conditions — Cystic Fibrosis; Digestive System Diseases; Genetic Diseases, Inborn; Lung Diseases; Pancreatic Diseases; Pathologic Processes; Respiratory Tract Diseases | interventions — Saline Solution, Hypertonic; Control Groups; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment Group (Experimental): 7% Hypertonic Saline administered via inhalation twice daily for 48 weeks
  Interventions: Drug: Active Treatment Group 7% Hypertonic Saline
- Control Group (Active Comparator): 0.9% Isotonic Saline administered via inhalation twice daily for 48 weeks
  Interventions: Drug: Control Group 0.9% Isotonic Saline

INTERVENTIONS:
Drug: Active Treatment Group 7% Hypertonic Saline — Drug: 7% Hypertonic Saline (HS) 4 mL of HS will be administered via inhalation twice daily for 48 weeks. The delivery system is a PARI Sprint Junior nebulizer with a PARI Baby face mask or mouthpiece driven by a PARI compressor (PARI Vios® Pro in USA, PARI BOY SX in Australia and Europe).
  Other Names:
  Hyper-Sal™, inhaled saline
  Arms: Active Treatment Group
Drug: Control Group 0.9% Isotonic Saline — Drug: 0.9% Isotonic Saline (IS) 4 mL of IS will be administered via inhalation twice daily for 48 weeks The delivery system is the same as that for the test product.
  Other Names: Normal saline
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess whether inhalation of 7% hypertonic saline (HS) twice daily for 48 weeks reduces structural lung disease as assessed by computed tomography (CT) in comparison with inhalation of 0.9% isotonic saline (IS) in preschool children (ages 3 to 6) with cystic fibrosis.

DETAILED DESCRIPTION:
Several observational studies have shown that cystic fibrosis (CF) patients less than or equal to 6 years of age have clinically silent airway damage. There is growing interest in early initiation of therapies to prevent or delay the progression of this lung disease in CF. In SHIP-CT, the investigators will evaluate treatment effects of HS relative to IS on measures of structural lung disease obtained from chest CT using a novel scoring system sensitive to early lung changes, the Perth-Rotterdam Annotated Grid Morphometric Analysis method for CF (PRAGMA-CF), that quantifies the volume percentage of diseased airways (%Dis), bronchiectasis (%Bx), and trapped air (%TA). As a secondary evaluation of structural airway damage, the investigators will use an image analysis system to measure airway dimensions relative to adjacent arteries (AA-system). Longitudinal changes in CT measures will also be compared to changes in lung function measured by the lung clearance index (LCI) obtained by N2 Multiple Breath Washout (MBW) and to clinical outcomes.

The primary hypothesis is that HS will reduce structural lung disease as assessed by the PRAGMA-CF computed tomography score relative to IS during the 48-week treatment period among preschool children with CF.

SHIP-CT is a parallel study to SHIP001 (ClinicalTrials.gov Identifier NCT02378467). The primary hypothesis of SHIP001, which runs in North America, is that compared to IS, HS will improve the LCI, a measure of ventilation heterogeneity, during the 48-week treatment period among preschool children with CF. The SHIP-CT study (SHIP002) will use a nearly identical study design as the SHIP001 study, with similar eligibility criteria and treatment arms, to determine whether HS reduces structural lung disease as measured by chest computed tomography (CT), in addition to stabilizing or improving functional outcomes as measured by LCI.

This is a multicenter, randomized, double-blind, controlled, parallel group trial assessing structural lung disease in children with CF ages 3 to 5 at enrollment. Participants will be randomized 1:1 to receive 7% hypertonic saline (treatment arm) vs. 0.9% isotonic saline (control arm) administered twice daily via jet nebulizer for 48 weeks. Study visits will occur at screening, enrollment, and at Weeks 12, 24, 36, and 48. Parents or the legal guardian will be contacted at Weeks 1, 4 and 8 to document changes in health status, adverse events, concomitant medications/treatments, and encourage study treatment compliance. Parents or the legal guardian will also be contacted approximately every 6 weeks between visit 3, 4, 5, and 6 to address individual issues or concerns related to study treatment or study participation, and to document changes in health status, medications and treatments.

Total duration of participant participation will be up to 53 weeks. As enrollment will occur over approximately 18 months, total duration of the study is expected to be up to 30 months (18 months enrollment plus 12 months for the last participants to complete study participation).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF as evidenced by one or more clinical features consistent with the CF phenotype or positive CF newborn screen AND one or more of the following criteria:

   1. A documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis (QPIT)
   2. A documented genotype with two disease-causing mutations in the CFTR gene
2. Informed consent by parent or legal guardian
3. Age ≥ 36 months and ≤72 months at screening visit
4. Ability to comply with medication use, study visits and study procedures as judged by the site investigator
5. Ability to cooperate with chest CT at the enrollment visit as determined by the lung function technician

Exclusion Criteria:

1. Chest CT within 8 months prior to the Screening visit
2. Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset within 3 weeks preceding screening or enrollment visit
3. Acute wheezing at screening or enrollment visit
4. Oxygen saturation < 95% (<90% in centers located above 4000 feet elevation) at screening or enrollment visit
5. Other major organ dysfunction, excluding pancreatic dysfunction
6. Physical findings that would compromise the safety of the participant or the quality of the study data as determined by site investigator
7. Investigational drug use within 30 days prior to screening or enrollment visit
8. Treatment with inhaled HS at any concentration within 30 days prior to screening or enrollment visit
9. Initiation (i.e. new prescription) of any inhaled hydrating agent such as mannitol or mucolytic agents such as dornase alpha within 30 days prior to the screening or enrollment visit
10. Chronic lung disease not related to CF
11. Inability to tolerate first dose of study treatment at the enrollment visit

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Chest CT | 48 weeks
  The difference in PRAGMA-CF %Dis between HS and IS study arm at end of study (48 weeks), adjusted for baseline, measured from standardized chest CT.

SECONDARY OUTCOMES:
PRAGMA-CF Sub-scores | 48 weeks
  i) The difference in PRAGMA-CF sub-scores, %Bx (the volume proportion of the lung with bronchiectasis) and %TA (the volume proportion of the lung with trapped air), between the baseline CT and the 48 week CT.
  ii) The absolute number of airways, airway dimensions and AA ratios from TLC CTs, acquired at the 48-week visit.
Lung Clearance Index (LCI) | 48 weeks
  The difference in LCI, measured by N2 MBW, from baseline to 48 weeks
Cross-sectional and longitudinal relationships | 48 weeks
  Cross-sectional and longitudinal relationships between primary and secondary PRAGMA-CF outcomes (%Dis, %Bx and %TA) and MBW outcomes (LCI), airway dimensions and PRAGMA-CF and MBW outcomes, as well as CFQ-R scores and PRAGMA-CF and MBW

CONTACTS AND LOCATIONS:
Overall Officials: Harm Tiddens, MD, PhD, Principal Investigator — Erasmus Medical Centre, Rotterdam; Stephen Stick, MD, PhD, Principal Investigator — Telethon Kids Institute, Perth; Margaret Rosenfeld, MD, MPH, Principal Investigator — Seattle Children's Hospital, Seattle; Stephanie Davis, MD, Principal Investigator — Indiana University, Indianapolis; Felix Ratjen, MD, PhD, FRCPC, Principal Investigator — The Hospital for Sick Children
Locations (25):
- United States (7):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Riley Hospital for Children, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Australia (7):
  - Royal Women's and Children Hospital, Adelaide
  - Lady Cilento Children's Hospital, Brisbane
  - Royal Children's Hospital, Melbourne
  - John Hunter Children's Hospital, Newcastle
  - Children's Hospital at Westmead, Sydney
  - Sydney Children's Hospital at Randwick, Sydney
  - Perth Children's Hospital, West Perth
- Belgium (2):
  - Universitair Ziekenhuis Children's Hospital, Brussels
  - UZ Leuven - Gasthuisberg Ziekenhuis, Leuven
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Kids, Toronto, Ontario
- Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Hospice Civils de Lyon, Lyon
  - Hospital Robert Debre, Paris
- Italy (2):
  - Bambini Gesu Children's Hospital, Roma
  - Ospedale Civile Maggiore, Verona
- Sophia Children's Hospital at Erasmus Medical Centre, Rotterdam, Netherlands
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenow T, Oudraad MC, Murray CP, Turkovic L, Kuo W, de Bruijne M, Ranganathan SC, Tiddens HA, Stick SM; Australian Respiratory Early Surveillance Team for Cystic Fibrosis (AREST CF). PRAGMA-CF. A Quantitative Structural Lung Disease Computed Tomography Outcome in Young Children with Cystic Fibrosis. Am J Respir Crit Care Med. 2015 May 15;191(10):1158-65. doi: 10.1164/rccm.201501-0061OC. PMID 25756857
- [Background] Ramsey KA, Rosenow T, Turkovic L, Skoric B, Banton G, Adams AM, Simpson SJ, Murray C, Ranganathan SC, Stick SM, Hall GL; AREST CF. Lung Clearance Index and Structural Lung Disease on Computed Tomography in Early Cystic Fibrosis. Am J Respir Crit Care Med. 2016 Jan 1;193(1):60-7. doi: 10.1164/rccm.201507-1409OC. PMID 26359952
- [Result] Tiddens HAWM, Chen Y, Andrinopoulou ER, Davis SD, Rosenfeld M, Ratjen F, Kronmal RA, Hinckley Stukovsky KD, Dasiewicz A, Stick SM; SHIP-CT Study Group. The effect of inhaled hypertonic saline on lung structure in children aged 3-6 years with cystic fibrosis (SHIP-CT): a multicentre, randomised, double-blind, controlled trial. Lancet Respir Med. 2022 Jul;10(7):669-678. doi: 10.1016/S2213-2600(21)00546-4. Epub 2022 Mar 11. PMID 35286860
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35286860/